CLINICAL TRIAL: NCT04335994
Title: ENhancing Outcomes in Cognitive Impairment Through Use of Home Sleep ApNea Testing: A Randomized Controlled Trial (ENCHANT Study)
Brief Title: ENhancing Outcomes in Cognitive Impairment Through Use of Home Sleep ApNea Testing
Acronym: ENCHANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 090-2019
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea; Alzheimer Disease; Vascular Dementia; Mild Cognitive Impairment; Parkinsons Disease With Dementia; Dementia With Lewy Bodies; Mixed Dementia
Keywords: Obstructive Sleep Apnea; Cognitive Impairment; Home Sleep Apnea Test; Screening
MeSH Terms: conditions — Sleep Apnea, Obstructive; Alzheimer Disease; Dementia, Vascular; Cognitive Dysfunction; Lewy Body Disease; Mixed Dementias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Patients receive standard of care for diagnosing obstructive sleep apnea, which is in-laboratory polysomnography.
  Interventions: Device: In-laboratory polysomnography
- Home Sleep Apnea Test (Experimental): Patients will undergo assessment for obstructive sleep apnea using a home sleep apnea test.
  Interventions: Device: Home Sleep Apnea Test

INTERVENTIONS:
Device: In-laboratory polysomnography — Level 1 in-laboratory polysomnography for the detection of obstructive sleep apnea.
  Other Names: iPSG
  Arms: Standard of Care
Device: Home Sleep Apnea Test — Use of a home sleep apnea test that records respiratory effort, pulse, oxygen saturation and nasal flow, and reports apneas, hypopneas, flow limitation, snoring and blood oxygen saturation in order to detect obstructive sleep apnea.
  Other Names: HSAT
  Arms: Home Sleep Apnea Test

SUMMARY:
Obstructive sleep apnea (OSA), which causes abnormal pauses in breathing during sleep, is common in patients with vascular cognitive impairment (VCI) and Alzheimer's disease (AD), and exacerbates the cognitive deficits seen in these conditions. OSA is typically treated with continuous positive airway pressure (CPAP), which has been shown to improve cognition in VCI and slow cognitive decline in AD. Despite the need to identify OSA in patients with VCI/AD, these patients often do not undergo testing for OSA. One major barrier is that in-laboratory polysomnography (iPSG), the current standard for diagnosing OSA, is inconvenient for patients with VCI/AD who may be reliant on others for care or require familiar sleep environments. A convenient and cheaper alternative to iPSG is home sleep apnea testing (HSAT), which has been validated against iPSG to diagnose OSA and has proven feasible for use in VCI/AD. Our primary objective is to determine whether the use of HSAT is superior to iPSG in terms of the proportion of patients who complete sleep testing by 6 months post-randomization. We will also investigate cost-effectiveness, patient satisfaction, proportion of patients treated with CPAP, changes in cognition, mood, sleep-related and functional outcomes between HSAT and iPSG at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of cognitive impairment by any one of: (i) Montreal Cognitive Assessment (MoCA) score of 13-28, or (ii) Mini Mental State Examination (MMSE) score of 18-30, or (iii) Toronto Cognitive Assessment (TorCA) score ≤281.
* A diagnosis of: (i) Single-domain amnestic or multiple cognitive domain (with one feature being amnestic) Mild Cognitive Impairment due to Alzheimer's disease (AD); or (ii) Probable AD dementia; or (iii) Possible AD dementia due to limited concomitant cerebrovascular disease; or (iv) Probable Vascular dementia or Vascular Mild Cognitive Impairment, as per the 2011 American Heart Association Scientific Statement; or (v) Patients with a suspected neurodegenerative condition known to be associated with non-OSA sleep disorders (e.g. Parkinson's disease-related dementia and dementia with Lewy Bodies); and/or (vi) Mixed disease
* Have the competency to provide informed consent, or the availability of a substitute decision maker/caregiver who can provide consent (if needed).
* The availability of a caregiver to assist in the completion of HSAT or iPSG, if needed.

Exclusion Criteria:

* Prior diagnosis of OSA within the last 2 years
* Patients already using CPAP or a dental appliance for previously diagnosed OSA.
* A known contraindication for the use of the HSAT that will be used in this study: (a) Moderate to severe pulmonary disease or congestive heart failure that could compromise the validity of the HSAT results (in users of the ApneaLink); (b) Permanent pacemaker or history of sustained non-sinus cardiac arrhythmia (in users of the WatchPAT).
* Any medical device that would interfere with the placement of the HSAT
* Significant physical impairment or language barrier that would restrict the ability to use the HSAT or complete the study assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete sleep testing | 6 months
  Proportion of patients who complete sleep testing by 6 months

SECONDARY OUTCOMES:
Proportion of patients diagnosed with OSA and treated using CPAP | 6 months
  Proportion of patients diagnosed with OSA and treated using CPAP by 6 months
Cognitive Outcomes (as assessed by the Montreal Cognitive Assessment) | 6 months
  Cognitive Outcomes (as assessed by the Montreal Cognitive Assessment) at 6 months
Cognitive Outcomes (as assessed by the Psychomotor Vigilance Task) | 6 months
  Cognitive Outcomes (as assessed by the Psychomotor Vigilance Task) at 6 months
Sleep-related quality of life (as assessed by the Functional Outcomes of Sleep Questionnaire) | 6 months
  Sleep-related quality of life (as assessed by the Functional Outcomes of Sleep Questionnaire) at 6 months
Mood (as assessed by the Geriatric Depression Scale) | 6 months
  Mood (as assessed by the Geriatric Depression Scale) at 6 months
Daytime Sleepiness (as assessed by the Epworth Sleepiness Scale) | 6 months
  Daytime Sleepiness (as assessed by the Epworth Sleepiness Scale) at 6 months
Health Related Quality of Life (as assessed by the EQ-5D-5L) | 6 months
  Health Related Quality of Life (as assessed by the EQ-5D-5L) at 6 months
Patient satisfaction for each strategy and treatment (as assessed by a Likert scale) | 6 months
  Patient satisfaction for each strategy and treatment (as assessed by a Likert scale) at 6 months
Cost to deliver each management strategy and treatment | 6 months
  Cost to deliver each management strategy and treatment by 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark I Boulos, MD, MSc, Principal Investigator — University of Toronto and Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No